CLINICAL TRIAL: NCT01050673
Title: A Study to Investigate the Time to Closure of Delayed Healing Dehisced Incisions, Delayed Healing Traumatic Wounds or Chronic Cutaneous Defects Surgically Excised With VERSAJET Compared Conventional Operating Room Techniques
Brief Title: Trial of Versajet Compared With Conventional Treatment in Acute and Chronic Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE/030/VJT
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Results first posted 2012-10-08 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Surgical Wound Dehiscence
Keywords: VERSAJET hydro-surgical debridement; traumatic wound
MeSH Terms: conditions — Surgical Wound Dehiscence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VERSAJET (Active Comparator): Excision with VERSAJET™ Hydrosurgery System
  Interventions: Device: VERSAJET
- Conventional Therapy (Active Comparator): Conventional operating room excision will consist of sharp instrumentation and electrocautery techniques, with the use of pulse lavage at the investigator's discretion. The type of sharp instrumentation, together with the brand of pulse lavage will be recorded.
  Interventions: Procedure: Scalpel or blade

INTERVENTIONS:
Device: VERSAJET — Hydro-surgery debridement
  Arms: VERSAJET
Procedure: Scalpel or blade — Conventional Surgical Debridement
  Arms: Conventional Therapy

SUMMARY:
It is increasingly recognised that the debridement of devitalised, bacterially contaminated or senescent tissue is an essential component of the effective treatment of delayed healing wounds.

Whilst surgical debridement procedures have conventionally been performed with scalpels and other sharp instrumentation, alternative techniques such as the VERSAJET Hydrosurgery System are becoming more widespread.

To increase the adoption of this new technology, it is essential that clinical improvements are assessed alongside the potential impact on the costs of debridement and the net financial impact on the hospital.

It is hypothesised that a decrease in the time to achieve stable wound closure will not only lead to a patient benefit, but also a potential reduction in the cost of treatment due to e.g. repeat procedures, longer hospital stay, infection etc. The purpose of this study is to investigate the difference in time to closure of wounds surgically excised with VERSAJET Hydrosurgery System and those surgically excised using conventional operating room techniques.

DETAILED DESCRIPTION:
It is increasingly recognised that the debridement of devitalised, bacterially contaminated or senescent tissue is an essential component of the effective treatment of delayed healing wounds. Whilst passive autolytic or enzymatic debridement procedures have their place, where patients are unable to tolerate any surgical procedure, the judicious use of surgical debridement to rapidly remove necrotic, contaminated tissue and slough has been shown to offer many advantages in returning a wound to a healing trajectory.

Whilst surgical debridement procedures have conventionally been performed with scalpels and other sharp instrumentation, alternative techniques such as the VERSAJET Hydrosurgery System are becoming more widespread.

To increase the adoption of this new technology, it is essential that clinical improvements are assessed alongside the potential impact on the costs of debridement and the net financial impact on the hospital. In fiscal year 2004, there were more than 57,000 discharges under DRG code 217 ('wound debridement and skin graft except hand) in the United States. Mean length of stay (all payers) was 11 days and mean charges were $52,800. In 2005, Medicare funded 15,800 discharges under this code. Average charges for these patients were $56,500 and average reimbursement was $18,2654. In this context it is particularly important that the potential patient benefit and cost impact of new technology is fully assessed.

It is hypothesised that a decrease in the time to achieve stable wound closure will not only lead to a patient benefit, but also a potential reduction in the cost of treatment due to e.g. repeat procedures, longer hospital stay, infection etc. The purpose of this study is to investigate the difference in time to closure of wounds surgically excised with VERSAJET Hydrosurgery System and those surgically excised using conventional operating room techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Male, and female patients (provided they are not pregnant and if of reproductive age are using contraception)
* Patients with a delayed healing traumatic wound or chronic cutaneous defect of 30 days or more in duration, or a delayed healing dehisced incision that requires excision to remove necrotic or infected tissue
* Patients who are deemed to require closure by primary intention or definitive cover with an autologous split-thickness skin graft (STSG) or flap
* Patients who are hospital in-patients, or will be an in-patient for the period of 1st excision to closure
* Patients deemed suitable for debridement with both VERSAJET Hydrosurgery System and conventional operating room techniques
* Patients undergoing surgical excision of their reference wound in the operating room (OR)
* Patients able to understand the evaluation and willing to consent to the evaluation

Exclusion Criteria:

* Patients who have previously undergone surgical excision of the reference wound by the Principal Investigator in the last 30 days
* Patients with coagulopathy (including those with haemophilia)
* Patients with vasculitis, non-reconstructive peripheral vascular disease, pyoderma granulosa, renal failure or lymphoedema
* Patients with irradiated, burn or ischaemic wounds
* Patients with a BMI >35
* Patients deemed to require a staged procedure, with hospital discharge occurring between procedures
* Patients deemed to require biological dressings / skin substitutes
* Patients for whom wound healing by secondary intention is deemed necessary
* Patients who have been treated with systemic immunosuppressants (including corticosteroids), or cytotoxic chemotherapy in the last 30 days, or who are anticipated to require such medications during the course of the study
* Patients known to have Acquired Immunodeficiency Syndrome (AIDS) or known to be infected with Human Immunodeficiency Virus (HIV)
* Patients with a known history of poor compliance with medical treatment
* Patients who have participated in this evaluation previously or who are currently participating in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-11; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Galiano, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

REFERENCES:
- [Background] Attinger CE, Janis JE, Steinberg J, Schwartz J, Al-Attar A, Couch K. Clinical approach to wounds: debridement and wound bed preparation including the use of dressings and wound-healing adjuvants. Plast Reconstr Surg. 2006 Jun;117(7 Suppl):72S-109S. doi: 10.1097/01.prs.0000225470.42514.8f. PMID 16799376
- [Background] Steed DL, Donohoe D, Webster MW, Lindsley L. Effect of extensive debridement and treatment on the healing of diabetic foot ulcers. Diabetic Ulcer Study Group. J Am Coll Surg. 1996 Jul;183(1):61-4. PMID 8673309

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VERSAJET | Conventional Therapy
Started | 21 | 19
Completed | 17 | 14
Not Completed | 4 | 5
Not completed — Physician Decision | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VERSAJET | Conventional Therapy | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 19 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (15.5) | 57.1 (13.7) | 54.5 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 16 | 10 | 26
Region of Enrollment [Number; unit: participants]
  United States | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Difference in Time to Closure Between Wounds Surgically Excised With VERSAJET™ Hydrosurgery System and Those Surgically Excised Using Conventional Operating Room Techniques.
Time Frame: 28 days plus 6 week follow-up
Measure: Median (Standard Deviation); unit: Time (minutes)
Arm/Group | VERSAJET | Conventional Therapy
Number analyzed (Participants) | 21 | 19
Time (minutes) | 7 (3.7) | 15 (8.5)

2. Secondary Outcome: Time of Actual Excision Procedure
Time Frame: 28 days
Measure: Median (Standard Deviation); unit: Time (Minutes)
Arm/Group | VERSAJET | Conventional Therapy
Number analyzed (Participants) | 21 | 19
Time (Minutes) | 7 (3.7) | 15 (8.5)

3. Secondary Outcome: Cost Per Operative Procedure
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: Dollars $
Arm/Group | VERSAJET | Conventional Therapy
Number analyzed (Participants) | 21 | 19
Dollars $ | 4411.70 (2020.2) | 6014.10 (4143.3)

4. Secondary Outcome: Cost of Reference Wound-related Surgical Procedures to Achieve Closure
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: Dollars ($)
Arm/Group | VERSAJET | Conventional Therapy
Number analyzed (Participants) | 21 | 19
Dollars ($) | 13689.1 (8154.3) | 12869.4 (5703.3)

5. Secondary Outcome: Quantitative Bacteriology From Standardised Tissue Biopsies Pre- /Post- 1st Excision & Pre-closure
Time Frame: 28 days
Population: Pre and post-excision values added, (cfu/g) tissue.
Measure: Median (Standard Deviation); unit: cfu/g
Arm/Group | VERSAJET | Conventional Therapy
Number analyzed (Participants) | 20 | 19
cfu/g
  Pre-first excision bacterial count (log10) cfu/g | 4.0 (2.1) | 4.0 (1.5)
  Post-first excision bacterial count (log10) cfu/g | 3.2 (2.0) | 3.3 (1.6)

6. Secondary Outcome: Percentage of Patients Achieving Stable Closure Within Study Period
Time Frame: 28 days
Measure: Number; unit: percentage of patients
Arm/Group | VERSAJET | Conventional Therapy
Number analyzed (Participants) | 21 | 19
percentage of patients | 42.9 | 42.1

7. Secondary Outcome: Length of Hospital Stay (1st Excision to Discharge (Days))
Time Frame: 28 days
Measure: Median (Standard Deviation); unit: Days
Arm/Group | VERSAJET | Conventional Therapy
Number analyzed (Participants) | 21 | 17
Days | 39 (22.6) | 38 (18.7)

8. Secondary Outcome: Number of Patient's With Wound-related Readmissions
Time Frame: 28 days and 6 week follow up
Measure: Number; unit: Number of patients
Arm/Group | VERSAJET | Conventional Therapy
Number analyzed (Participants) | 21 | 19
Number of patients | 1 | 0

9. Secondary Outcome: Number of Patient's With Serious Adverse Events and Relationship to Device
Time Frame: 28 days
Measure: Number; unit: Number of patients
Arm/Group | VERSAJET | Conventional Therapy
Number analyzed (Participants) | 21 | 19
Number of patients | 5 | 5

ADVERSE EVENTS:
Arm/Group | VERSAJET | Conventional Therapy
Serious Adverse Events (participants affected / at risk) | 5/21 | 5/19
Other Adverse Events (participants affected / at risk) | 0/21 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VERSAJET (N=21) | Conventional Therapy (N=19)
calcaneal pin site infection leading to foot gangrene (Infections and infestations) | 1 (1) | 0 (0)
sacral pressure sore (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
urinary tract infection (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
flap dehiscence (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
flap failure (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
seroma leading to limited flap dehiscence (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
infection leading to prolonged hospitalisation and an amputation of the distal portion of the right (Infections and infestations) | 0 (0) | 1 (1)
partial flap failure/dehiscence (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No